CLINICAL TRIAL: NCT02833285
Title: Periodontitis and Inflammation : Biological and Clinical Approach of B Cell Role.
Brief Title: B Cell Functions in Periodontitis
Acronym: LBPARO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: LBPARO
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-05

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — gingiva biopsy gingival fluid blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The inflammatory response involves many players from the immune response, including B lymphocytes. These cells are responsible for the synthesis of immunoglobulins in response to the presence of an antigen. They are characteristic of chronic inflammation. There are several subsets of B cells characterized by specific membrane markers. Once activated, these cells express many factors contributing to tissue destruction seen in periodontitis and particularly in osteoclastogenesis (receptor activator of nuclear factor kappa-B ligand, tumor necrosis factor, interleukin-6, macrophage inflammatory protein-1α and Monocyte Chemoattractant Protein-3).

During the establishment of a periodontal disease, an important inflammatory infiltrate is observed in the gum. This infiltrate is characterized by the presence of many B lymphocytes. B cell subsets in the blood and the gum of patients with periodontitis have been little studied. However, the number of autoreactive B cells (cluster of differentiation (CD)19+, CD5+) has been reported to be higher in the blood of patients with periodontal disease. In the gum, the rate of B and T cells increases with the level of inflammation and is correlated with the severity of the inflammatory process. Activation of B cells is a prerequisite for the progression of gingivitis to periodontitis. B cell distribution could then be an indicator of disease progression, but also allow to study the response to treatment.

The aim of this pilot study is to characterize B cell subsets in the blood and the gum of patients with periodontitis, according to disease activity. Analysis of B cells in the blood could highlight the association of a particular subpopulation with aggressive periodontal disease and evidence a particular biological profile of the host response. The investigators also wish to observe the evolution of this phenotype following an unconventional surgical therapy.

This study would better understand the pathogenesis of periodontal disease and refine the diagnosis, prognosis and treatment of periodontitis, and thus participate in the development of personalized medicine. Biological monitoring of therapeutic effects may be initiated and allow more effectively prevent recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Requiring periodontal surgery
* In good health
* Having signed consent

Exclusion Criteria:

* Minor
* Patient having taken antibiotics in the previous 3 months
* Patients with systemic diseases including chronic inflammatory disease
* Pregnancy
* orthodontic treatment ongoing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female from 18 to 75 years old before periodontal treatment
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Phenotype of B cells in the blood and gums | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: ALARD Jean-Eric, Principal Investigator — University Hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demoersman J, Pochard P, Framery C, Simon Q, Boisrame S, Soueidan A, Pers JO. B cell subset distribution is altered in patients with severe periodontitis. PLoS One. 2018 Feb 15;13(2):e0192986. doi: 10.1371/journal.pone.0192986. eCollection 2018. PMID 29447240